CLINICAL TRIAL: NCT03579498
Title: Brain Function After Cardiac Arrest (Measured With FMRI and Cognitive Tests)
Acronym: BRAINnHEART
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Sten Rubertsson, Professor Anaesthesiology & Intensive Care Medicine, Uppsala University
Other Study IDs: BH001
Record Dates: First submitted 2018-05-17; First posted 2018-07-06 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Cardiac Arrest; Cognitive Function
Keywords: Cardiac arrest; Cognitive impairment; Depression; Anxiety; PTSD; Health- related quality of life; functional MRI
MeSH Terms: conditions — Heart Arrest; Cognitive Dysfunction; Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: Patients who have suffered a cardiac arrest at Uppsala University Hospital or who were admitted to this hospital after the event.
- Control group: The control group will, as far as it is possible, match the patient group regarding mean age, age distribution, sex and educational attainments.

SUMMARY:
The aim of this longitudinal study is to determine whether brain function is affected after a cardiac arrest.

The primary question is whether cognitive function is affected after cardiac arrest and whether it changes over time (during the first year after the event), compared with a healthy control group. Brain function during cognitive tasks and emotion processing will also be studied using functional MRI (fMRI). Another aim is to study whether clinical outcomes such as PTSD, anxiety and depression can be correlated with cognitive function and whether health- related quality of life is affected after a cardiac arrest.

The results from the cardiac arrest patient group will be compared with a healthy control group.

DETAILED DESCRIPTION:
The study is a prospective cohort study and aims to enroll 30 cardiac arrest patients and 30 matched (regarding age, gender and level of education), healthy controls.

Patients who are enrolled in the study will on three different occasions (in the acute phase, after six and after twelve months) answer questions regarding their health state and perform a computerized cognitive test and a behavioral test.

Patient/ control health status will be assessed through the following tests:

* Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCa) screening tool which measures attention/concentration, executive functions, memory, verbal skills, visual construction skills, abstract thinking, computation and orientation.
* Presence of delirium will be assessed using the Confusion Assessment Method for the Intensive Care Unit (CAM- ICU) and will be complemented with information from the patients' medical records.
* The Richmond Agitation - Sedation Scale (RASS) will be used to assess sedation.
* Health- related quality of life will be measured using the three level version of EQ-5D (EQ-5D-3L; Euro-Qol 5-Dimensions).
* A Mini International Neuropsychiatric Interview (MINI) will be performed to detect psychiatric syndromes (such as PTSD, anxiety and depression). Symptoms of anxiety and depression will also be measured using The Montgomery-Åsberg Depression Rating Scale- Self report (MADRS-S) and Impact of Event Scale-Revised -22. Alcohol use will be assessed using AUDIT (Alcohol Use Disorders Identification Test).

Information will also be collected from the patients' medical records.

Cognitive/ neuropsychological testing will be performed using the Cambridge Neuropsychological Test Automated Battery (CANTAB), which measures amongst others memory, planning, executive functions and attention. For this study, the following CANTAB modules will be used:

* Delayed matching to sample (DMS)
* Paired associate learning test (PAL)
* Stockings of Cambridge (SOC)/ One Touch Stockings of Cambridge (OTS)
* Motor Screening Task (MOT), which provides a general assessment of whether sensorimotor deficits or lack of comprehension will limit the collection of valid data from the participant.

The tests are performed on a tablet. All task stimuli are non- verbal.

An approach- avoidance test that measures avoidance behavior will also be performed. Patients will be presented with auditory and visual (pictures) stimuli and will choose whether the stimuli presented to them will be of a neutral or aversive character. Patients will be informed that choosing the aversive stimuli will reward them with a small amount of money.

Functional magnetic resonance imaging (fMRI) will be performed six and twelve months after the cardiac arrest. The MRI scan will also include morphological images. The fMRI sequence will include tests regarding emotional activation, emotional memory and cognitive interference. A DMS task with emotionally loaded stimuli will be performed. Blood oxygenation level dependent (BOLD)- imaging will be used to produce the fMRI images, where differences in blood flow in different parts of the brain will be registered through echo planar imaging (EPI). The images will be analyzed with the Statistical Parametric Mapping (SPM)-12 program using MATLAB computing language.

The healthy control group will on two occasions (with the second occasion taking place six months after the first) answer questions regarding their health state, perform cognitive testing and fMRI. The same will be assessed for the control as for the patient group, with the exception of CAM-ICU, RASS and information from medical records, which will not be included in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have suffered a cardiac arrest of cardiac cause who were admitted to hospital after the event.
* Age 18-70
* Consents to participating in the study

Exclusion Criteria:

* Terminal disease with expected survival <1 year, moribund patient with >1 treatment limitations.
* A history of brain injury or brain disease that affects cognitive function, such as dementia
* Severe psychiatric disorder, for example psychotic disorders or severe alcohol use disorder
* Insufficient knowledge of the spoken language to understand instructions and answer questionnaires (oral or written)
* Deceased within 1 month.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 30 cardiac arrest patients and 30 matched (regarding age, gender and educational level), healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Cognitive function after cardiac arrest and changes over time | 2-6 weeks, 6 and 12 months post- cardiac arrest
  Cognitive function in cardiac arrest survivors according to CANTAB and MoCa. Measured in the acute phase (2-6 weeks), 6 and 12 months post- cardiac arrest. Comparison with healthy controls

SECONDARY OUTCOMES:
Health- related quality of life after cardiac arrest | 2-6 weeks, 6 and 12 months post- cardiac arrest
  Health- related quality of life according to the three level (3L) version of Euro-Qol 5-Dimensions (5D), EQ-5D-3L, which consists of a descriptive system and a visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self- care, usual activities, pain/discomfort and anxiety/depression. Each dimension has three levels from which the subject chooses the most appropriate statement : 1 (no problems), 2 (some problems) and 3 (extreme problems). The results are calculated as an index, ranging from -0,594 (death, or worse than death) to 1 (full health), based on normative data in the population. The EQ VAS is a scale where subjects rate their health from 0 (labeled "The worst health you can imagine) and 100 (labeled "The best health you can imagine).
  Measured in the acute phase (2-6 weeks), 6 and 12 months post- cardiac arrest. Comparison with healthy controls and correlation with depression, anxiety, PTSD and cognitive function.
Depression after cardiac arrest according to MINI- interviews | 2-6 weeks, 6 and 12 months post- cardiac arrest
  Prevalence of depression according to MINI- interviews. Measured in the acute phase (2-6 weeks), 6 and 12 months post- cardiac arrest. Comparison with healthy controls and correlation with cognitive function and health- related quality of life.
Depression after cardiac arrest according to MADRS-S | 2-6 weeks, 6 and 12 months post- cardiac arrest
  Prevalence of depression according to MADRS-S. The scale measures depressive symptoms and consists of nine items (mood, feelings of unease, sleep, appetite, ability to concentrate, initiative, emotional involvement, pessimism and zest for life). Each item has seven levels (0-6, where higher scores indicate increased impairment) with described statements from which the subject chooses the most appropriate statement. The total score is then calculated as a sum of the individual scores. The total score ranges from 0 to 60 points and is interpreted as follows: 0-12 points: no depression/ essentially unaffected; 13-19 points: mild depression; 20-34 points: moderate depression; >34 points: severe depression.
  Measured in the acute phase (2-6 weeks), 6 and 12 months post- cardiac arrest. Comparison with healthy controls and correlation with cognitive function and health- related quality of life.
Anxiety after cardiac arrest | 2-6 weeks, 6 and 12 months post- cardiac arrest
  Prevalence of anxiety according to MINI- interviews. Measured in the acute phase (2-6 weeks), 6 and 12 months post- cardiac arrest. Comparison with healthy controls and correlation with cognitive function and health- related quality of life.
PTSD after cardiac arrest | 2-6 weeks, 6 and 12 months post- cardiac arrest
  Prevalence of post- traumatic stress syndrome (PTSD) according to MINI- interviews. Measured in the acute phase (2-6 weeks), 6 and 12 months post- cardiac arrest. Comparison with healthy controls and correlation with cognitive function and health- related quality of life.
Return to daily functioning after cardiac arrest according to questionnaires and interviews | 2-6 weeks, 6 and 12 months post- cardiac arrest
  Return to daily functioning in cardiac arrest survivors. In the acute phase (2-6 weeks) patients report current and previous (prior to the cardiac arrest) occupation and living arrangements. The same questions, as well as an interview regarding self- perceived return to daily life, will be answered at 6 and 12 months after the cardiac arrest. Return to daily functioning is defined as return to the same level of independence, living arrangements, occupation, family life, social interactions as well as engagement in leisure activities as prior to the cardiac arrest.
Prevalence of neuroanatomical deficits after cardiac arrest | 6 months post- cardiac arrest
  Prevalence of neuroanatomical deficits, such as infarcts, after cardiac arrest. Visualized by first MRI (6 months post- cardiac arrest). Comparison with healthy controls.
Change in affective and cognitive processing, regional reactivity and connectivity measured through fMRI after cardiac arrest | 6 and 12 months post- cardiac arrest
  Change in affective and cognitive processing, regional reactivity and connectivity after cardiac arrest. Changes in regional oxygen consumption and blood flow during a DMS task with emotionally loaded stimuli will be assessed through fMRI. fMRI will be performed 6 and 12 months post- cardiac arrest. Comparison with healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rubertsson, Prof, MD, Principal Investigator — Uppsala University Hospital
Locations (2):
- Haukeland University Hospital, Bergen, Norway
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Background] Buanes EA, Gramstad A, Sovig KK, Hufthammer KO, Flaatten H, Husby T, Langorgen J, Heltne JK. Cognitive function and health-related quality of life four years after cardiac arrest. Resuscitation. 2015 Apr;89:13-8. doi: 10.1016/j.resuscitation.2014.12.021. Epub 2015 Jan 14. PMID 25596374
- [Background] Bush G, Shin LM, Holmes J, Rosen BR, Vogt BA. The Multi-Source Interference Task: validation study with fMRI in individual subjects. Mol Psychiatry. 2003 Jan;8(1):60-70. doi: 10.1038/sj.mp.4001217. PMID 12556909
- [Background] Cunningham JL, Wernroth L, von Knorring L, Berglund L, Ekselius L. Agreement between physicians' and patients' ratings on the Montgomery-Asberg Depression Rating Scale. J Affect Disord. 2011 Dec;135(1-3):148-53. doi: 10.1016/j.jad.2011.07.005. PMID 21856017
- [Background] Hariri AR, Mattay VS, Tessitore A, Kolachana B, Fera F, Goldman D, Egan MF, Weinberger DR. Serotonin transporter genetic variation and the response of the human amygdala. Science. 2002 Jul 19;297(5580):400-3. doi: 10.1126/science.1071829. PMID 12130784
- [Background] Larsson C, Axell AG, Ersson A. Confusion assessment method for the intensive care unit (CAM-ICU): translation, retranslation and validation into Swedish intensive care settings. Acta Anaesthesiol Scand. 2007 Aug;51(7):888-92. doi: 10.1111/j.1399-6576.2007.01340.x. PMID 17635396
- [Background] Larsson IM, Wallin E, Rubertsson S, Kristofferzon ML. Health-related quality of life improves during the first six months after cardiac arrest and hypothermia treatment. Resuscitation. 2014 Feb;85(2):215-20. doi: 10.1016/j.resuscitation.2013.09.017. Epub 2013 Oct 2. PMID 24096198
- [Background] Larsson IM, Wallin E, Rubertsson S, Kristoferzon ML. Relatives' experiences during the next of kin's hospital stay after surviving cardiac arrest and therapeutic hypothermia. Eur J Cardiovasc Nurs. 2013 Aug;12(4):353-9. doi: 10.1177/1474515112459618. Epub 2012 Sep 14. PMID 22984190
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Reinert DF, Allen JP. The Alcohol Use Disorders Identification Test (AUDIT): a review of recent research. Alcohol Clin Exp Res. 2002 Feb;26(2):272-9. PMID 11964568
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Sveen J, Orwelius L, Gerdin B, Huss F, Sjoberg F, Willebrand M. Psychometric properties of the Impact of Event Scale-Revised in patients one year after burn injury. J Burn Care Res. 2010 Mar-Apr;31(2):310-8. doi: 10.1097/BCR.0b013e3181d0f523. PMID 20182373
- [Background] Torgersen J, Hole JF, Kvale R, Wentzel-Larsen T, Flaatten H. Cognitive impairments after critical illness. Acta Anaesthesiol Scand. 2011 Oct;55(9):1044-51. doi: 10.1111/j.1399-6576.2011.02500.x. Epub 2011 Sep 8. PMID 22092200
- See also: The EuroQol database — http://www.euroqol.org/